CLINICAL TRIAL: NCT04670042
Title: Feasibility and Effectiveness of Using Peripheral Nerve Stimulation (PNS) to Treat Chronic Post-surgical Pain (CPSP) Following Total Knee Arthroplasty.
Brief Title: Using Peripheral Nerve Stimulation (PNS) to Treat Chronic Post-surgical Pain (CPSP) After Knee Surgery
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Difficulty enrolling in this patient population
Sponsor: Stanford University (Other)
Collaborators: SPR Therapeutics, Inc. (Industry)
Responsible Party: Principal Investigator, Einar Ottestad, Clinical Associate Professor, Stanford University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 58819
Record Dates: First submitted 2020-11-11; First posted 2020-12-17 (Actual); Last update posted 2022-10-20 (Actual); Status verified 2022-10

CONDITIONS: Injury; Nerve, Peripheral, Multiple; Chronic Post-Procedural Pain; Total Knee Arthroplasty; Surgery; Knee Injuries; Knee Pain Chronic; Postoperative Pain; Chronic Postoperative Pain
Keywords: Chronic Pain Following Left Total Knee Arthroplasty; Chronic Pain Following Right Total Knee Arthroplasty
MeSH Terms: conditions — Wounds and Injuries; Knee Injuries; Pain, Postoperative | interventions — Drug Delivery Systems

STUDY DESIGN:
Intervention Model Description: Case series of 15 subjects with chronic post-surgical pain (CPSP). Subjects will be recruited over 6 months (on average 1 subject per week)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (1):
- SPRINT® Peripheral Nerve Stimulation (PNS) System (Experimental): SPRINT PNS System will be offered to patients with postoperative knee pain following primary unilateral total knee arthroplasty (TKA) who meet eligibility criteria and consistent with established coverage policy. SPRINT PNS System will be implanted for 60 days. At the discretion of the physician, the first lead may be placed to stimulate the nerve innervating the region of greatest pain. If pain is not adequately addressed by the first lead when assessed at 10 days, a second lead may be placed approximately 2 weeks following the initial lead placement.
  Interventions: Device: SPRINT® Peripheral Nerve Stimulation (PNS) System (510k Cleared)

INTERVENTIONS:
Device: SPRINT® Peripheral Nerve Stimulation (PNS) System (510k Cleared) — Same as Arm Description.

SUMMARY:
SPRINT PNS System will be offered to patients with postoperative knee pain following primary unilateral total knee arthroplasty (TKA) who meet eligibility criteria and consistent with established coverage policy. SPRINT PNS System will be implanted for 60 days. At the discretion of the physician, the first lead may be placed to stimulate the nerve innervating the region of greatest pain. If pain is not adequately addressed by the first lead when assessed at 10 days, a second lead may be placed approximately 2 weeks following the initial lead placement.

ELIGIBILITY:
Inclusion Criteria:

* At least 21 years old
* Underwent a primary or revision unilateral TKA
* Completed all CHOIR questionnaires before and after TKA surgery
* Persistent postsurgical knee pain ≥ 5 of 10 during ambulation as demonstrated on the CHOIR assessment.
* Must meet the definition of chronic pain.

  1. Pain that continues or is expected to continue for longer than 3 months from its initial onset or
  2. Persistent pain that at the discretion of the physician has not resolved within the normal time course of healing or
  3. Pain requiring opioid use beyond 30 days.

Exclusion Criteria:

* Patients with a pre-operative history of moderate to high dose use of opioids (≥ 50 morphine milligram equivalents (MME) average per day)
* Patients taking opioids for reasons other than pain in knee that underwent TKA
* Patients with arthrofibrosis or indicated for manipulation under anesthesia
* BMI >35
* Uncontrolled Diabetes Mellitus Types I or II, indicated by an HbA1c >7.0% within the last 3 months
* Vulnerable population (e.g. pregnant women, prisoners, minors, or employees)
* Deep brain stimulation (DBS) system, an implanted active cardiac implant, or any other implantable neurostimulator whose stimulus current pathway may overlap the SPRINT stimulator's current pathway.
* Any other condition that may interfere with the ability to participate in a clinical trial (e.g., anatomy that may interfere with lead placement, nerve damage in affected leg, pain caused by knee implant requiring revision, compromised immune system) as determined by the Investigator
* Workers Compensation

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2021-06-25 (Actual); Primary Completion 2022-08 (Estimated); Study Completion 2024-05 (Estimated)

PRIMARY OUTCOMES:
Change in Pain Intensity from Baseline to 12 Months | Collected at baseline, 10, 30, 60, and 90 days post lead placement; and 6 months following TKA
  The primary outcome is Pain Intensity using Numerical Rating Scale (NRS) from 0-10 with the higher number (10) being worse pain and (0) being no pain.
  Incidence of chronic post-surgical pain (CPSP) through Pain Intensity will be looked at for patients throughout the study along with usage of the Peripheral Nerve Stimulation (PNS) device (hours/day).
  A collection of surveys already approved for patients following total knee arthroplasty from Stanford's Collaborative Health Outcomes Information Registry (CHOIR) will also be sent to patients.

SECONDARY OUTCOMES:
Change in Opioid Use | Collected at baseline, 10, 30, 60, and 90 days post lead placement; and 6 months following TKA
  Opioid use as documented in the medical records and patient-reported.
  Will note the increase, decrease, or no change in opioid associated with implantation of the study device.

CONTACTS AND LOCATIONS:
Overall Officials: Einar Ottestad, Principal Investigator — CLINICAL ASSOCIATE PROFESSOR, ANESTHESIOLOGY, PERIOPERATIVE AND PAIN MEDICINE
Locations (1):
- Stanford Pain Management Center, Redwood City, California, United States

IPD SHARING:
Plan to Share IPD: No
Not Sharing.

REFERENCES:
- [Background] Gilmore C, Ilfeld B, Rosenow J, Li S, Desai M, Hunter C, Rauck R, Kapural L, Nader A, Mak J, Cohen S, Crosby N, Boggs J. Percutaneous peripheral nerve stimulation for the treatment of chronic neuropathic postamputation pain: a multicenter, randomized, placebo-controlled trial. Reg Anesth Pain Med. 2019 Jun;44(6):637-645. doi: 10.1136/rapm-2018-100109. Epub 2019 Apr 5. PMID 30954936
- [Background] Ilfeld BM, Said ET, Finneran JJ 4th, Sztain JF, Abramson WB, Gabriel RA, Khatibi B, Swisher MW, Jaeger P, Covey DC, Robertson CM. Ultrasound-Guided Percutaneous Peripheral Nerve Stimulation: Neuromodulation of the Femoral Nerve for Postoperative Analgesia Following Ambulatory Anterior Cruciate Ligament Reconstruction: A Proof of Concept Study. Neuromodulation. 2019 Jul;22(5):621-629. doi: 10.1111/ner.12851. Epub 2018 Aug 30. PMID 30160335
- [Background] Ilfeld BM, Gabriel RA, Said ET, Monahan AM, Sztain JF, Abramson WB, Khatibi B, Finneran JJ 4th, Jaeger PT, Schwartz AK, Ahmed SS. Ultrasound-Guided Percutaneous Peripheral Nerve Stimulation: Neuromodulation of the Sciatic Nerve for Postoperative Analgesia Following Ambulatory Foot Surgery, a Proof-of-Concept Study. Reg Anesth Pain Med. 2018 Aug;43(6):580-589. doi: 10.1097/AAP.0000000000000819. PMID 29905630
- [Background] Ilfeld BM, Gilmore CA, Grant SA, Bolognesi MP, Del Gaizo DJ, Wongsarnpigoon A, Boggs JW. Ultrasound-guided percutaneous peripheral nerve stimulation for analgesia following total knee arthroplasty: a prospective feasibility study. J Orthop Surg Res. 2017 Jan 13;12(1):4. doi: 10.1186/s13018-016-0506-7. PMID 28086940
- [Background] Ilfeld BM, Ball ST, Gabriel RA, Sztain JF, Monahan AM, Abramson WB, Khatibi B, Said ET, Parekh J, Grant SA, Wongsarnpigoon A, Boggs JW. A Feasibility Study of Percutaneous Peripheral Nerve Stimulation for the Treatment of Postoperative Pain Following Total Knee Arthroplasty. Neuromodulation. 2019 Jul;22(5):653-660. doi: 10.1111/ner.12790. Epub 2018 Jul 19. PMID 30024078
- See also: Peripheral Nerve Stimulator Device Website — https://www.sprtherapeutics.com/